CLINICAL TRIAL: NCT02254460
Title: A Double Blind, Randomized, Two-way Cross-over Study to Investigate the Uptake of Iron From Micronutrient Fortified Powder vs. From Tailored Control in Milk.
Brief Title: Investigation of Iron Uptake From Micronutrient Fortified Powder Versus From Tailored Control in Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 202738; RH01592 (Other: GSK)
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Growth and Development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Experimental product: Micronutrient fortified beverage powder, packed as 27 g individual sachet, administered orally as a single serve.
  Interventions: Dietary Supplement: Test
- Control (Placebo Comparator): Energy equivalent beverage powder without micronutrient fortification, packed as 27 g individual sachets, administered orally as a single serve
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Test — Experimental product: Micronutrient fortified beverage powder, packed as 27 g individual sachet, administered orally as a single serve.
  Arms: Test
Other: Control — Energy equivalent beverage powder without micronutrient fortification, packed as 27 g individual sachets, administered orally as a single serve
  Arms: Control

SUMMARY:
The present study supplements iron as part of multiple micro-nutrient supplementation to demonstrate that intake of a micronutrient fortified powder in milk helps increase the uptake of key micronutrients like iron due to unique nature of the given matrix, as compared to intake of iron alone in milk.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study and willingness to participate as evidenced by participants' parents and/or legal guardian's voluntary written informed consent as well as written assent by the participant and has received a signed and dated copy of the informed consent form as well as the assent form
* Participant belonging to middle socio-economic background as per modified Kuppuswamy scale
* Good general and mental health with, in the opinion of the investigator or medically qualified designee
* Child residing in the peri-urban areas of Bangalore city
* Child with Z-scores of: a. height for age of 0 to ≥-3; b. BMI for age of 0 to ≥-3.

Exclusion Criteria:

* Children in Care (CiC)
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds), any of their stated ingredients or any known food allergies like peanut allergy, gluten allergy or lactose intolerance
* Participants with severe anaemia (Haemoglobin < 8g %) as determined by laboratory results
* Current or relevant history of any serious, severe or unstable physical or psychiatric illness or any medical disorder that would make the participant unlikely to fully complete the study or any condition that presents undue risk from the study product or procedures in the opinion of the investigator
* Recent history (3 months) of serious infections, injuries and/ or surgeries
* Children consuming iron, calcium and/or other nutritional supplements and/ or health food drinks on a regular basis (more than 3 times a week) in last 6 months prior to screening visit
* Use of any prescription medications within 15 days prior to screening and throughout the entire duration of the study
* Recent history (within the last 1 year) of alcohol or other substance abuse.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2013-02-06; Primary Completion 2013-03-01 (Actual); Study Completion 2013-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bangalore, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from two centers in India.
Pre-assignment Details: A total of 37 participants were screened, 25 were randomized and 24 completed the study. One participant withdrew from the study due to an adverse event (AE).
Groups:
- Test Followed by Control: Patients first received micronutrient fortified nutritional beverage powder (test) and then energy, iron and calcium equivalent beverage powder without micronutrient fortification (control), packed as 27 grams (g) individual sachets, administered as a single serve in a total volume of 100 milliliters (mL) lukewarm milk for oral consumption. 1mL solution containing 3 milligrams/milliliters (mg/mL) of the stable iron isotope (57Fe,58Fe) was added to the graduated drinking container followed by a sachet of the study beverage powder. Lukewarm milk was added to the container to make up the volume to 100mL of reconstituted beverage
- Control Follwed by Test: Patients first received energy, iron and calcium equivalent beverage powder without micronutrient fortification (control) and then micronutrient fortified nutritional beverage powder (test), packed as 27g individual sachets, administered as a single serve in a total volume of 100mL of lukewarm milk for oral consumption. 1mL solution containing 3mg/mL of the stable iron isotope (57Fe,58Fe) was added to the graduated drinking container followed by a sachet of the study beverage powder. Lukewarm milk was added to the container to make up the volume to 100mL of reconstituted beverage.
Period: Overall Study
Arm/Group | Test Followed by Control | Control Follwed by Test
Started | 13 | 12
Completed | 12 | 12
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: Micronutrient fortified nutritional beverage powder (test) and energy, iron and calcium equivalent beverage powder without micronutrient fortification (control), packed as 27 g individual sachets, administered as a single serve in a total volume of 100 mL lukewarm milk for oral consumption. 1mL solution containing 3mg/mL of the stable isotope (57Fe,58Fe) was added to the graduated drinking container followed by a sachet of the study beverage powder. Lukewarm milk was added to the container to make up the volume to 100mL of reconstituted beverage.
Arm/Group | Overall
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Years | 8.60 (1.000)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Fractional Iron Absorption
Description: Iron uptake was measured using stable isotopes of 57Fe and 58Fe to label the test and control products. Fractional iron absorption levels of 57Fe and 58Fe were calculated, to give a direct measure of the iron uptake from each of the study treatments.
Time Frame: Day 15
Population: Per protocol (PP) population, defined as all participants who received at least one study treatment administration and who did not have any protocol violations deemed to affect evaluation of the iron absorption. This analysis was conducted on PP population.
Measure: Mean (Standard Deviation); unit: % Iron Absorbed
Groups:
- Test: Micronutrient fortified nutritional beverage powder, packed as 27g individual sachets, administered as a single serve in a total volume of 100 mL lukewarm milk for oral consumption. 1mL solution containing 3mg/mL of the stable iron isotope (57Fe,58Fe) was added to the graduated drinking container followed by a sachet of the study beverage powder (test). Lukewarm milk was added to the container to make up the volume to 100mL of reconstituted beverage.
- Control: Energy, iron and calcium equivalent beverage powder without micronutrient fortification, packed as 27g individual sachets, administered as a single serve in a total volume of 100mL of lukewarm milk for oral consumption.1mL solution containing 3mg/mL of the stable iron isotope (57Fe,58Fe) was added to the graduated drinking container followed by a sachet of the study beverage powder (control). Lukewarm milk was added to the container to make up the volume to 100mL of reconstituted beverage.
Arm/Group | Test | Control
Number analyzed (Participants) | 24 | 24
% Iron Absorbed | 2.08 (1.263) | 1.25 (0.922)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Superiority or Other; p = 0.0944, ANOVA; [Treatment difference] = 1.74, 95% CI 2-sided [0.90 to 3.34] — Treatment difference from ANOVA of log transformed data. Back transformed data are presented. This therefore represents the iron absorption ratio of the Micronutrient Fortified Drink (Test) to the Non-Fortified Drink (Control)

ADVERSE EVENTS:
Groups:
- Control: Energy, iron and calcium equivalent beverage powder without micronutrient fortification, packed as 27g individual sachets, administered as a single serve in a total volume of 100mL of lukewarm milk for oral consumption. 1mL solution containing 3mg/mL of the stable iron isotope (57Fe, 58Fe) was added to the graduated drinking container followed by a sachet of the study beverage powder (control). Lukewarm milk was added to the container to make up the volume to 100mL of reconstituted beverage.
Arm/Group | Test | Control
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 1/25 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test (N=25) | Control (N=24)
Gastritis (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.